CLINICAL TRIAL: NCT01231867
Title: Clopidogrel and Proton Pump Inhibitors: A Propensity Score Adjusted Cohort Study to Examine a Possible Interaction: A CALIBER Study
Brief Title: Cohort Study of Clopidogrel and Proton Pump Inhibitors
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Ian Douglas, Senior Lecturer, London School of Hygiene and Tropical Medicine
Other Study IDs: 09_042; CALIBER 09_09
Record Dates: First submitted 2010-10-18; First posted 2010-11-01 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Heart Disease; Acute Coronary Syndrome; Drug Interactions; Clopidogrel; Proton Pump Inhibitors; Gastrointestinal Hemorrhage
Keywords: Coronary Heart Disease; Acute Coronary Syndrome; Drug interactions; Clopidogrel; Proton Pump Inhibitors; Gastrointestinal Hemorrhage
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients who have experienced and survived non-ST segment elevation acute coronary syndromes are often prescribed a combination of aspirin and clopidogrel to thin the blood and prevent further acute coronary episodes. Both clopidogrel and aspirin may cause stomach bleeds and so a prophylactic proton pump inhibitor is frequently co-prescribed in order to prevent such bleeds. Recent mechanistic and observational studies suggest proton pump inhibitors may reduce the effectiveness of clopidogrel and so patients may not benefit as much as expected from combined aspirin and clopidogrel. The investigators propose a cohort study of patients prescribed clopidogrel + aspirin. Amongst these patients the investigators will measure the relative rate of acute coronary syndrome and death comparing patients with and without proton pump inhibitor treatment. To provide a more complete picture of the risks and benefits of treatment the investigators will also measure the relative rate of stomach bleeds in the same groups of patients. In addition, whether the inhibitory effect of proton pump inhibitors on the protective effect of clopidogrel is due to their inhibition of drug metabolising enzymes will be explored by assessing the effects of other drugs that inhibit the same enzymes.

DETAILED DESCRIPTION:
Background

Patients who have experienced and survived non-ST segment elevation acute coronary syndromes are often prescribed a combination of aspirin and clopidogrel to thin the blood and prevent further acute coronary episodes. Both clopidogrel and aspirin may cause stomach bleeds and so a prophylactic proton pump inhibitor is frequently co-prescribed in order to prevent such bleeds. Recent mechanistic and observational studies suggest proton pump inhibitors may reduce the effectiveness of clopidogrel and so patients may not benefit as much as expected from combined aspirin and clopidogrel. The investigators propose a cohort study of patients prescribed clopidogrel + aspirin. Amongst these patients the investigators will measure the relative rate of acute coronary syndrome and death comparing patients with and without proton pump inhibitor treatment. To provide a more complete picture of the risks and benefits of treatment the investigators will also measure the relative rate of stomach bleeds in the same groups of patients. In addition, whether the inhibitory effect of proton pump inhibitors on the protective effect of clopidogrel is due to their inhibition of drug metabolising enzymes will be explored by assessing the effects of other drugs that inhibit the same enzymes.

Background Clopidogrel is an antiplatelet drug used to prevent coronary events, particularly in patients who have already experienced acute coronary syndrome (ACS). It is often used in combination with aspirin, and due to the propensity of both drugs to cause gastrointestinal (GI) bleeds, prophylactic therapy with proton pump inhibitor (PPI) is frequently prescribed. Some proton pump inhibitors and clopidogrel share a common metabolic pathway involving the cytochrome P450 2C19 isoenzyme. Clopidogrel relies on P450 2C19 for conversion to its active metabolite whilst some PPIs inhibit this enzyme; recent mechanistic studies suggest that PPIs may reduce the platelet inhibitory effect of clopidogrel (Gilard et al 2006, Gilard et al 2008). Subsequent observational studies appear to show this effect may translate directly to a reduction in clopidogrel efficacy with patients more likely to experience secondary coronary events or death. Odds ratios of 1.25 (95% confidence interval (CI) 1.11-1.41; Ho et al 2009) and 1.27 (1.03-1.57; Juurlink et al 2009) have been reported, comparing clopidogrel and PPI users with patients using clopidogrel without PPI. A further study suggests the effect may be limited to clopidogrel in combination with omeprazole only (Sibbing et al 2009).

Scientific hypothesis

Main Research Questions: To investigate a possible drug interaction between clopidogrel and proton pump inhibitors (PPI). Specific questions to be answered are:

1. Does combined use of clopidogrel/aspirin with a PPI increase the risk of acute coronary syndrome or death compared with clopidogrel/aspirin without a PPI, and if so by how much?
2. Does combined use of clopidogrel/aspirin with a PPI decrease the risk of gastrointestinal bleed compared with clopidogrel/aspirin without a PPI and if so by how much?

Objectives

Using the cohort method we will:

1. Estimate the rate ratio for acute coronary syndrome or death, comparing individuals prescribed clopidogrel + aspirin with a PPI with individuals prescribed clopidogrel + aspirin without a PPI.
2. Estimate the rate ratio for gastrointestinal bleed, comparing individuals prescribed clopidogrel + aspirin with a PPI with individuals prescribed clopidogrel + aspirin without a PPI.
3. Estimate the rate ratio for acute coronary syndrome or death, comparing individuals prescribed clopidogrel + aspirin with non-PPI cytochrome P450 2C19 inhibitors with individuals prescribed clopidogrel + aspirin without non-PPI cytochrome P450 2C19 inhibitors using the cohort method

Methodology and planned statistical analyses A cohort study is proposed to address the issues outlined above. This is the optimum design since it will allow us to measure relative and absolute rates of the events of interest. We will also be able to assign follow up time to different exposure groups as dictated by patient prescriptions.

Study Population: All patients registered in the General Practice Research Database (GPRD) from 1998 to date and receiving clopidogrel in combination with aspirin and with at least 12 months up-to-standard observation before the first prescription for clopidogrel will be eligible for inclusion. Data will be restricted to 1998 onwards as this is the year clopidogrel was licensed in the United Kingdom (UK).

Primary Exposure: Any PPI in combination with aspirin and clopidogrel. Prescriptions for PPI's, aspirin and clopidogrel will be identified from patient records.

Primary Outcome: A combined end point of all cause mortality OR incident myocardial infarction (MI). Mortality will be determined using the GPRD-estimated date of death and incident MI will be determined by searching clinical and referral records. Recent linkages between GPRD and the Myocardial Ischaemia National Audit Project [MINAP] will be exploited to validate event diagnoses and to ensure events are incident rather than prevalent (see sub-group analyses below).

Secondary Exposures: A combination of aspirin and clopidogrel with any of the following will be determined: CYP2C19 inhibiting PPIs, non-CYP2C19 inhibiting PPIs, omeprazole only, paroxetine or fluoxetine. Paroxetine and fluoxetine have been selected as they are CYP2C19 inhibitors likely to be widely used over long periods of time.

Secondary Outcomes: Incident GI bleed, incident MI.

Data Analysis: Data will be analysed using STATA v9.2 (StataCorp, Texas) using Cox regression and adjusting for possible confounders (see covariates below). Rate ratios (RR) and 95% confidence intervals will be estimated for the outcomes outlined above, comparing individuals exposed to aspirin + clopidogrel + PPI with people exposed to aspirin + clopidogrel + no PPI.

Follow up time for each individual will be classified according to the treatments being received at any point in time. We will use recorded data on dosing frequency and pack size to estimate the exposure period of each prescription. Where this data is missing, the median length of exposure calculated for all other prescriptions of that drug will be assumed.

Sub-group analyses: Since smoking is an important potential confounder and will not be recorded perfectly in the GPRD, sensitivity analyses will be undertaken. The main imprecision is likely to be among ex-smokers who are recorded as non-smokers. We will therefore undertake an analysis including only people recorded as definite "never smokers" and people recorded as current smokers.

Linkage between MINAP and GPRD is not available for all practices in the GPRD. All analyses using the MINAP-validated date of ACS event will be restricted to patients from practices where linkage has been established.

Sample Size and Power Calculation GPRD feasibility counts indicate >40,000 patients may have received clopidogrel and aspirin simultaneously and 31,000 of these have also received a PPI at some point. Assuming a study period incidence of the primary outcome of 25%1 and a conservative exposed/unexposed group size of 5,000 each, we would have >99% power to detect a rate ratio of 1.2 comparing the rate of death or MI among aspirin and clopidogrel users who are taking a PPI with those not taking a PPI. This would be consistent with the effect detected in studies to date (Ho et al 2009, Juurlink et al 2009).

Covariates

MI, mortality and GI bleeds have several well-established risk factors which are also likely to be associated with the exposures of interest in this study. We will therefore examine the possible confounding effects of the following covariates. The list includes covariates found to be associated with PPI treatment in the observational studies done in this area to date:

* Age, sex, general practice, smoking status, alcohol consumption, body mass index
* History of:- diabetes, MI, percutaneous coronary intervention, coronary artery bypass graft surgery, heart failure, cerebrovascular disease, cancer, chronic obstructive pulmonary disease, renal disease, hepatic disease, dementia, GI bleed, peripheral vascular disease, other atherosclerotic disease.

It is possible that some patients receiving clopidogrel + aspirin with a PPI will differ from those not prescribed a PPI to such an extent that comparisons of the rate of MI, mortality and GI bleeds may be invalid. To investigate this possibility we will calculate propensity scores for PPI treatment using baseline characteristics. Only patients with propensity scores within a common range between the 2 groups will be included in the cohort analysis, ensuring a fair comparison.

This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD), secondary care (HES) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset)

ELIGIBILITY:
Inclusion Criteria:

* All patients registered in the GPRD from 1998 to date and receiving clopidogrel in combination with aspirin and with at least 12 months up to standard observation before the first prescription for clopidogrel will be eligible for inclusion

Exclusion Criteria:

* Data will be restricted to 1998 onwards as this is the year clopidogrel was licensed in the UK.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients registered in the GPRD from 1998 to date and receiving clopidogrel in combination with aspirin and with at least 12 months up to standard observation before the first prescription for clopidogrel will be eligible for inclusion. Data will be restricted to 1998 onwards as this is the year clopidogrel was licensed in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 24471 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Time to composite end point of all cause mortality OR incident myocardial infarction (MI) | up to 12 years

SECONDARY OUTCOMES:
Time to incident gastrointestinal (GI) bleed. | up to 12 years
Time to incident myocardial infarction | up to 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Douglas, PhD, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- London School of Hygiene & Tropical Medicine, London, United Kingdom

REFERENCES:
- [Background] Gilard M, Arnaud B, Le Gal G, Abgrall JF, Boschat J. Influence of omeprazol on the antiplatelet action of clopidogrel associated to aspirin. J Thromb Haemost. 2006 Nov;4(11):2508-9. doi: 10.1111/j.1538-7836.2006.02162.x. Epub 2006 Aug 8. No abstract available. PMID 16898956
- [Background] Gilard M, Arnaud B, Cornily JC, Le Gal G, Lacut K, Le Calvez G, Mansourati J, Mottier D, Abgrall JF, Boschat J. Influence of omeprazole on the antiplatelet action of clopidogrel associated with aspirin: the randomized, double-blind OCLA (Omeprazole CLopidogrel Aspirin) study. J Am Coll Cardiol. 2008 Jan 22;51(3):256-60. doi: 10.1016/j.jacc.2007.06.064. PMID 18206732
- [Background] Ho PM, Peterson ED, Wang L, Magid DJ, Fihn SD, Larsen GC, Jesse RA, Rumsfeld JS. Incidence of death and acute myocardial infarction associated with stopping clopidogrel after acute coronary syndrome. JAMA. 2008 Feb 6;299(5):532-9. doi: 10.1001/jama.299.5.532. PMID 18252883
- [Background] Juurlink DN, Gomes T, Ko DT, Szmitko PE, Austin PC, Tu JV, Henry DA, Kopp A, Mamdani MM. A population-based study of the drug interaction between proton pump inhibitors and clopidogrel. CMAJ. 2009 Mar 31;180(7):713-8. doi: 10.1503/cmaj.082001. Epub 2009 Jan 28. PMID 19176635
- [Background] Sibbing D, Morath T, Stegherr J, Braun S, Vogt W, Hadamitzky M, Schomig A, Kastrati A, von Beckerath N. Impact of proton pump inhibitors on the antiplatelet effects of clopidogrel. Thromb Haemost. 2009 Apr;101(4):714-9. PMID 19350116
- [Derived] Douglas IJ, Evans SJ, Hingorani AD, Grosso AM, Timmis A, Hemingway H, Smeeth L. Clopidogrel and interaction with proton pump inhibitors: comparison between cohort and within person study designs. BMJ. 2012 Jul 10;345:e4388. doi: 10.1136/bmj.e4388. PMID 22782731
- See also: General Practice Research Database — http://gprd.com
- See also: CALIBER — http://www.caliberresearch.org